CLINICAL TRIAL: NCT00001008
Title: Pharmacokinetic Study of the Interaction of Azidothymidine and Methadone in Patients With AIDS and ARC
Brief Title: A Study of Azidothymidine Plus Methadone in Patients With AIDS and AIDS Related Complex (ARC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 055
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 1991-08

CONDITIONS: HIV Infections
Keywords: Substance Withdrawal Syndrome; Methadone; Opioid-Related Disorders; Drug Evaluation; Drug Interactions; Drug Therapy, Combination; Administration, Oral; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Substance Withdrawal Syndrome; Opioid-Related Disorders; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Methadone; Zidovudine

INTERVENTIONS:
Drug: Methadone hydrochloride
Drug: Zidovudine

SUMMARY:
To determine if methadone treatment will affect the blood levels of zidovudine (AZT) in patients with AIDS or AIDS-related complex (ARC) who are receiving oral AZT and methadone therapy. In addition, the blood levels of methadone both before and during AZT treatment will be studied, and patients receiving daily oral methadone treatment will be evaluated for signs of narcotic withdrawal during treatment with AZT.

The number of deaths due to AIDS in high-risk populations continues to increase. Nationwide approximately 25 percent of AIDS patients are intravenous (IV) drug abusers, and it is very likely that an increasingly larger number of AIDS patients receiving AZT therapy will have had a history of IV drug abuse. The major chemical treatment for IV drug abuse is daily methadone maintenance therapy, and IV drug abusers who are HIV positive represent a large number of patients who will undergo long-term treatment with both methadone and AZT. Therefore, the study of potential drug interactions is essential.

DETAILED DESCRIPTION:
The number of deaths due to AIDS in high-risk populations continues to increase. Nationwide approximately 25 percent of AIDS patients are intravenous (IV) drug abusers, and it is very likely that an increasingly larger number of AIDS patients receiving AZT therapy will have had a history of IV drug abuse. The major chemical treatment for IV drug abuse is daily methadone maintenance therapy, and IV drug abusers who are HIV positive represent a large number of patients who will undergo long-term treatment with both methadone and AZT. Therefore, the study of potential drug interactions is essential.

The 18 patients are patients with AIDS or ARC. Nine are control patients who are not receiving methadone and are not IV drug abusers. Nine are former IV drug abusers who have been maintained on methadone for at least 6 months and who have been receiving a constant daily dose of methadone for at least 1 month. Plasma and urine levels of methadone are determined over a 4 hour period. The dose of AZT: For the pharmacokinetic study of AZT, plasma and urine samples are taken after oral dose of AZT and an intravenous dose of AZT in the control and methadone groups.

ELIGIBILITY:
Inclusion Criteria

Prior Medication:

Allowed:

* Oral nonabsorbable antifungal agents.

The study will include 18 patients with AIDS or HIV-related symptomatic illness as defined by the CDC classification group IVa and c2. Of these, 9 methadone recipients will have been maintained on methadone for at least 1 month and will have received a constant daily dose of 30-90 mg of methadone for at least 10 days.

Nine patients will be former intravenous drug abusers.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Temperature > 101 degrees F.
* Ascites.
* Active opportunistic infection.

Concurrent Medication:

Excluded:

* Other inducers or inhibitors of hepatic microsomal enzymes.
* Any chronic systemic medications.

Patients with the following symptoms or conditions are excluded:

* Temperature > 101 degrees F.
* Ascites.
* Active opportunistic infection.

Prior Medication:

Excluded within 72 hours of study entry:

* All medication except oral nonabsorbable antifungal agents.
* Excluded within 2 weeks of study entry:
* Any other experimental drug.
* Drugs with known nephrotoxic potential or drugs known to cause neutropenia.
* Rifampin or its derivatives, phenytoin, or barbiturates.

Active drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Primary Completion 1991-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G Friedland, Study Chair
Locations (1):
- Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York, United States

REFERENCES:
- [Background] Schwartz EL, Brechbuhl AB, Kahl P, Miller MH, Selwyn PA, Friedland GH. Altered pharmacokinetics of zidovudine in former IV drug-using patients receiving methadone. Int Conf AIDS. 1990 Jun 20-23;6(3):194 (abstract no SB432)
- [Background] Schwartz EL, Brechbuhl AB, Kahl P, Miller MA, Selwyn PA, Friedland GH. Pharmacokinetic interactions of zidovudine and methadone in intravenous drug-using patients with HIV infection. J Acquir Immune Defic Syndr (1988). 1992;5(6):619-26. PMID 1588496